CLINICAL TRIAL: NCT00750711
Title: Typical Flutter Ablation:A Comparison of 4 mm Versus 2 mm Irrigated cathéters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Dipen Shah, University Hospital of Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocole 08-006
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2008-09-16 (Estimated); Status verified 2008-09

CONDITIONS: Typical Atrial Flutter; Radiofrequency Ablation; Irrigated Catheters
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KT,2 (Experimental): There are two arms in this study: KT2 arm and KT4 arm. Patients in KT2 arm will be ablated with the 2 mm irrigated catheter and patients in KT4 mm will be ablated with the 4 mm irrigated catheter.
  Interventions: Procedure: Radiofrequency ablation for atrial flutter by catheters

INTERVENTIONS:
Procedure: Radiofrequency ablation for atrial flutter by catheters

SUMMARY:
The purpose of this study is to compare the efficacy of 4 mm irrigated catheters with 2 mm irrigated catheters for ablation of typical flutter.It's a prospective randomised multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* All patients above the age 18 years undergoing a first catheter ablation for typical atrial flutter

Exclusion Criteria:

* Pregnancy
* Hemodynamic instability
* A recurrence of previous ablated typical atrial flutter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Procedural success rate, procedure duration, number of RF applications, delivered power, impedance, complication rate, recurrence at six months | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital of Geneva, Geneva, Canton of Geneva
  - University Hospital of Geneva, Geneva